CLINICAL TRIAL: NCT06203808
Title: Impact in Head and Neck Oncology of Support by a Nurse in the Patient's Care Pathway.
Acronym: COACH-ORL
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/23/0410
Record Dates: First submitted 2023-12-12; First posted 2024-01-12 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COACH GROUP: The COACH group consists of newly diagnosed head and neck cancer patients seen in consultation for treatment information at Oncologic University Hospital during the first two months of the study. These patients receive coaching support from a specialized nurse, facilitating appointment scheduling, treatment coordination, and access to various rehabilitation services
  Interventions: Other: COMPLETION OF QUESTIONNAIRES
- CONTROL GROUP: The control group includes patients who received the treatment information during the third and fourth months of the study, without receiving specific coaching support.
  Interventions: Other: COMPLETION OF QUESTIONNAIRES

INTERVENTIONS:
Other: COMPLETION OF QUESTIONNAIRES — Both groups of patients will complete quality of life questionnaires at the time of treatment information, at 3 months, 6 months and at 12 months.

SUMMARY:
Head and neck cancers (HNC) constitute a significant global health burden, ranking fourth in terms of cancer incidence and fifth in terms of cancer-related mortality. The management of HNC requires a complex array of consultations, examinations, rehabilitation, and lifestyle modifications, including addiction cessation. These cancers disproportionately affect economically disadvantaged, socially isolated individuals, and the elderly, resulting in disparities in healthcare access. Health coaching, an approach aimed at improving patients' health and quality of life by supporting behavior and lifestyle changes, has demonstrated effectiveness in various medical fields, including chronic diseases, medical oncology, and hematology. However, its application in head and neck cancer care remains limited, despite its potential benefits for this patient population.

DETAILED DESCRIPTION:
This study is a prospective monocentric comparative investigation conducted over 12 months. Two groups are being compared: the COACH group and the control group. The COACH group consists of newly diagnosed head and neck cancer patients seen in consultation for treatment information at University Hospital during the first two months of the study. These patients receive coaching support from a specialized nurse, facilitating appointment scheduling, treatment coordination, and access to various rehabilitation services. In contrast, the control group includes patients who received treatment information during the third and fourth months of the study, without receiving specific coaching support. Both groups of patients will complete quality of life questionnaires at the time of treatment information, at 3 months, 6 months, and at 12 months.

Hypothesis: the investigators assume a minimum difference of 5 points between the control group and the coaching group.

ELIGIBILITY:
Inclusion criteria:

* Patient with a histologically proven diagnosis of head and neck squamous cell carcinoma (HNSCC) of the upper aerodigestive tract
* Patient whose disease is classified UICC (Union for International Cancer Control (UICC) Tumour, Node, Metastasis (TNM) stage (8th edition): T0-4a NO/N3 M0 (no distant metastasis M0)
* Patient World Health Organization (WHO) 0-1-2
* Treatment with a feasible curative aim (no contraindication to optimal treatment such as surgery or chemotherapy at a curative dose)
* Patient affiliated to a Social Security scheme in France
* Patient who did not object to participating in the research.

Non-inclusion criteria:

* Patient with a history of previous cervical surgery and/or head and neck irradiation
* Pregnant or breastfeeding women
* Patient suffering from another co-existing malignant disease at the time of inclusion or any other significant medical (immunosuppression etc.), psychiatric or surgical condition, currently not controlled by treatment, which may interfere with the achievement of the study.
* Any psychological, family, geographic or sociological condition that does not allow compliance with medical monitoring and/or the procedures provided for in the study protocol.
* Patients deprived of liberty or under legal protection regime (curatorship and guardianship, safeguard of justice).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a histologically proven diagnosis of head and neck squamous cell carcinoma (HNSCC) of the upper aerodigestive tract
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Potential benefits of personalized patient support using European Organisation for Research and Treatment of Cancer (EORTC) questionnaire | 12 months
  The main objective of this study is to evaluate the impact on the quality of life of patients treated for upper aerodigestive tract cancer of support by a nurse during the care pathway; and this from the moment of diagnosis and up to 12 months afterwards.
  Measure of the impact on quality of life using the validated questionnaire most commonly used in oral cancerology, i.e. EORTC Quality of Life Questionnaire (QLQ) - Head and Neck Cancer (EORTC QLQ-H&N43).

CONTACTS AND LOCATIONS:
Overall Officials: AGNES DUPRET-BORIES, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Chu de Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided